CLINICAL TRIAL: NCT03875989
Title: Vaginal Native Tissues Repair for Pelvic Organ Prolapse
Acronym: TAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 87RI18_0013 (TAPP)
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Prolapse, Vaginal
Keywords: Prolapse; Vaginal native tissues repair; Pelvic organ
MeSH Terms: conditions — Uterine Prolapse; Prolapse

STUDY DESIGN:
Intervention Model Description: Experimental, parallel-group randomised controlled trial (1:1), multicentric. The primary outcome and the secondary outcome 1 and 3 will be evaluated in double blind; only the secondary outcome 2 will not be evaluated in blind.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator)
  Interventions: Procedure: Anterior colporraphy
- Arm B (Experimental)
  Interventions: Procedure: vaginal patch plastron

INTERVENTIONS:
Procedure: Anterior colporraphy — It will be delimitate a rectangular vaginal strip which will be isolated from the anterior colpocele. The superior edge of the strip is placed 2 cm from the urethral orifice. After lateral vesico-vaginal dissection, the paravesical fossae will be wide opened to repair the tendinous arches. The vaginal plastron will be fixed to the tendinous arch of the pelvic fascia by 3 lateral stitches (anterior/ lateral/ posterior) on each side of the plastron. After, the plastron will be tensioning and the cystocele will be suspended. The closure of the vaginal wall will end the procedure.
  Arms: Arm A
Procedure: vaginal patch plastron — It will be make a midline incision of the anterior vaginal wall from the urethrovesical junction to the vaginal apex or anterior fornix. The vaginal epithelium will be separated from the underlying fibromuscular layer (Halban Fascia) after the midline incision. Midline plication of the fibromuscular layer will be obtained by interrupted horizontal stiches. The closure of the vaginal wall will end the procedure.
  Arms: Arm B

SUMMARY:
The aim of the study is to assess at one year the effectiveness of the vaginal patch plastron in comparison of the anterior colporraphy through a combined definition of success: anatomic and functional.

DETAILED DESCRIPTION:
Pelvic organ prolapse is usually the result of loss of pelvic support. It is widely accepted that 50% of women after 50 years old will develop prolapse, evaluated through the POPQ Classification . Pelvic organ prolapse cause significant psychological distress and negatively affect quality of life. Among the surgery for prolapse, the cystocele cureis is the most frequent (67.7%). Native tissue cystocele repairs is the cornerstone of prolapse surgery especially since the learned societies (Food and Drug Administration, Haute Autorité de Santé, Collège National des Gynécologues-Obstétriciens Français) warned clinicians and patients about serious mesh related complications. In France, 41.5% of vaginal cystocele repair are with native tissue. The main surgeries are anterior colporraphy and vaginal patch plastron, used in routine in our center with re-intervention rates less than 4% at one year. Rate of success of native tissue cystocele repair are heterogeneous, depending on the design of studies and definition of outcomes. A prospective study find a success rate at 35% of the anterior colporraphy based on a combined definition, anatomic and functional as recommended recently. However the definition of anatomic was strict (POPQ<2), while it seems that the best definition of anatomic success is "no prolapse among the hymen", that is to say aAa and Ba points <0.

We think that the vaginal patch plastron will have a better anatomic and functional success comparatively to the anterior colporraphy as it corrects median cystoceles by a vaginal strip as well as lateral cystoceles by the bilateral paravaginal suspension.

The description of the two surgeries will be standardized between all the surgeons. We will compare the anterior colporraphy consisting in bladder median support by retensioning Halban fascia with colpectomy to the vaginal patch plastron consisting in making a vaginal strip attached to the bladder combined with suspension by fixation of the vaginal strip to the tendinous arch of the pelvic fascia.

Patients will be blind of their surgery. They will have a follow-up visit 45 days after the surgery to evaluate the post- operative complications according to the Clavien-Dindo classification. They will have phone call at 4 and 8 months after the surgery to make sure they've not suffered for complications. At last, they will have a follow-up visit 1 year after the surgery by an independent assessor blind of the surgery to evaluate the primary outcome (anatomic and functional success).

ELIGIBILITY:
Inclusion Criteria:

* Patient at 50 years of age or older
* Symptomatic primary prolapse of the anterior vaginal wall defined by Aa and/or Ba points ≥0 according to the POP-Q system
* A positive response to the question "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?" (question 3 of the PFDI-20)
* Able to give informed consent
* Performans Status score ≤ 2

Exclusion Criteria:

* Patient with need for surgical treatment for myorraphy of levator ani muscles
* Patient with previous surgical cystocele repair.
* Patient with evolving gynaecologic cancer.
* Pregnancy or wish for future pregnancy, lactating woman.
* Inability to participate in study follow-up or to provide informed consent.
* Lack of social insurance .

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2025-09-27 (Estimated); Study Completion 2028-03-27 (Estimated)

PRIMARY OUTCOMES:
Rate of the prolapse surgery | 1 year
  The success rate of the prolapse surgery defined by a composite of objective and subjective measures:
  * Anatomic success defined by Aa and Ba values <0 in Pelvic Organ Prolapse Quantification System (POP-Q) AND
  * Subjective success through reliable condition-specific quality-of-life questionnaires:
    * A negative response to the question "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?" (question 3 of the Pelvic Floor Distress Inventory (PFDI-20)) AND
    * Range score of Patient Global Impression of Improvement (PGI-I) 1 or 2 AND
  * No need for other treatment for prolapse (surgical nor medical)

SECONDARY OUTCOMES:
Rate of the prolapse surgery | 1 year
  The failure rate of the prolapse surgery defined by a composite of objective and subjective measures:
  * Recurrent prolapse defined by Aa and/or Ba values > or= 0 in POP-Q OR
  * Subjective failure through reliable condition-specific quality-of-life questionnaires:
    * A positive response to the question "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?" (question 3 of the PFDI-20) OR
    * A PGI-I score > 2 OR
  * Need of a new treatment for prolapse (surgical or medical)
Rate of post-operative complications | 45 Days
  Rate of post-operative complications according to the Clavien-Dindo classification 45 days after the surgery by the patient's surgeon (not blinded)
Sexual function | 1 year
  The sexual function improvement will be evaluated by the difference in PISQ 12 score (condition-specific quality-of-life questionnaire) between the inclusion and one year after the surgery for sexually active women
Rate of the prolapse surgery | 2 years
  The failure rate of the prolapse surgery defined by a composite of objective and subjective measures:
  * Recurrent prolapse defined by Aa and/or Ba values > or= 0 in POP-Q OR
  * Subjective failure through reliable condition-specific quality-of-life questionnaires:
    * A positive response to the question "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?" (question 3 of the PFDI-20) OR
    * A PGI-I score > 2 OR
  * Need of a new treatment for prolapse (surgical or medical)
Rate of the prolapse surgery | 3 years
  The failure rate of the prolapse surgery defined by a composite of objective and subjective measures:
  * Recurrent prolapse defined by Aa and/or Ba values > or= 0 in POP-Q OR
  * Subjective failure through reliable condition-specific quality-of-life questionnaires:
    * A positive response to the question "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?" (question 3 of the PFDI-20) OR
    * A PGI-I score > 2 OR
  * Need of a new treatment for prolapse (surgical or medical)

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU de Bordeaux, Bordeaux
  - CH de Brive, Brive-la-Gaillarde
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CH de Gueret, Guéret
  - CHU de Limoges, Limoges
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Toulouse - Paule de Viguier, Toulouse
  - CHU de Toulouse - Rangueil, Toulouse
  - CH de Tulle, Tulle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lacorre A, Vidal F, Campagne-Loiseau S, Marin B, Aubard Y, Siegerth F, Mesnard C, Chantalat E, Hocke C, Gauthier T. Protocol for a randomized controlled trial to assess two procedures of vaginal native tissue repair for pelvic organ prolapse at the time of the questioning on vaginal prosthesis: the TAPP trial. Trials. 2020 Jul 8;21(1):624. doi: 10.1186/s13063-020-04512-x. PMID 32641096